CLINICAL TRIAL: NCT03875391
Title: The Effect of Oxytocin on the Acquisition and Consolidation of Trauma-Associated Memories: A Model to Understand the Development of Posttraumatic Stress Disorder
Brief Title: The Effect of Oxytocin on the Consolidation of Trauma-Associated Memories
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Stefan Roepke, Principal Investigator, PD Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: Charite2019-Oxytocin-Study
Record Dates: First submitted 2019-03-11; First posted 2019-03-14 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2022-04

CONDITIONS: Intrusive Memories; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin and trauma film paradigm (Experimental): Intervention: Drug: Oxytocin nasal spray
  Interventions: Drug: Oxytocin
- Placebo and trauma film paradigm (Placebo Comparator): Intervention: Drug: Placebos
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Drug: Oxytocin nasal spray
  Arms: Oxytocin and trauma film paradigm
Drug: Placebo — Drug: Placebo nasal spray
  Arms: Placebo and trauma film paradigm

SUMMARY:
The purpose of the study is to examine whether oxytocin and certain polygenic risk scores affect the development of intrusive memories, a cardinal symptom of PTSD.

ELIGIBILITY:
Inclusion Criteria:

* healthy female volunteers
* German on a native level

Exclusion Criteria:

* former or present disorder according to the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5)
* any physical illnesses
* any medication intake (except oral contraceptive)
* history of traumatic experience, e.g. history of sexual abuse or rape
* pregnancy or lactation period
* follicular phase of menstrual cycle for all women not using oral contraceptives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change of Intrusive Memories in the following four days after the intervention | four consecutive days
  Influence of oxytocin on the development of intrusive memories measured with an intrusion diary

SECONDARY OUTCOMES:
Noradrenergic System (measured with salivary alpha-amylase - u/ml) | Day 1
  Influence of oxytocin on the noradrenergic system measured with salivary alpha-amylase
Hypothalamic-pituitary-adrenal (HPA) axis (measured with salivary cortisol - nmol/L) | Day 1
  Influence of oxytocin on the HPA-axis measured with salivary cortisol
Polygenic Risk Score | four consecutive days
  Influence of polygenic risk score on development of intrusive memories

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Roepke, Prof, Principal Investigator — Charité
Locations (1):
- Charité- Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Derived] Maslahati T, Wingenfeld K, Hellmann-Regen J, Kraft J, Lyu J, Keinert M, Voss A, Cho AB, Ripke S, Otte C, Schultebraucks K, Roepke S. Oxytocin vs. placebo effects on intrusive memory consolidation using a trauma film paradigm: a randomized, controlled experimental study in healthy women. Transl Psychiatry. 2023 Feb 4;13(1):42. doi: 10.1038/s41398-023-02339-z. PMID 36739422